CLINICAL TRIAL: NCT06375785
Title: Comparison of Two Different Exercise Methods in Geriatrics
Brief Title: Two Different Exercise Methods in Geriatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Collaborators: Fenerbahce University (Other); Istanbul Galata University (Other); Biruni University (Other)
Responsible Party: Principal Investigator, Gülsena Utku, Principal Investigator, Halic University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LSVT-BIG vs Otago
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Elderly People; Nursing Homes
Keywords: elderly people; LSVT-BIG; Otago; exercise; balance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Otago-based (slow rhythmic) exercise group (Experimental)
  Interventions: Other: Otago-based (slow rhythmic) exercise group
- Group 2 - LSVT BIG-based (large amplitude) exercise group (Experimental)
  Interventions: Other: LSVT BIG-based (large amplitude) exercise group

INTERVENTIONS:
Other: Otago-based (slow rhythmic) exercise group — Slow Rhythmic Exercises (Otago based) A.Strength training
  1. Knee flexion and extension
  2. Ankle dorsiflexion and plantar flexion
  3. Toes flexion and extension
  4. Hip abduction and adduction B. Balance training
  1. Stepping backwards, walking and turning 2.Side walking 3. Octet walking 4.Tandem walking 5. Standing up from a sitting position
  Arms: Group 1 - Otago-based (slow rhythmic) exercise group
Other: LSVT BIG-based (large amplitude) exercise group — Large Amplitude Exercises (based on LSVT-BIG)
  1. Bending towards the floor and rising towards the ceiling (opening) while sitting
  2. While sitting, turn to the right and left with the body and reach out
  3. Sit down
  4. Step forward
  5. Sidestepping
  6. Stepping back
  7. Step forward and extend arm towards the ceiling
  8. Step sideways and extend arm towards the ceiling
  9. Walking with big steps
  10. Turning from right to left and left to right while walking
  Arms: Group 2 - LSVT BIG-based (large amplitude) exercise group

SUMMARY:
The aim of the study is to compare slow rhythmic exercises with large amplitude exercises in elderly people

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older
* living in a nursing home
* Knowing how to read and write Turkish
* Cognitive functions are sufficient for communication (Standardized Mini Mental Test score over 21 points)
* Being between 1-5 on the Clinical Fragility Scale
* Not taking medical medications regularly due to pain
* Volunteering to participate in the study

Exclusion Criteria:

* Having vision and hearing problems that affect communication (except for individuals who communicate with glasses and hearing aids)
* Having a disease that causes neurological, orthopedic and musculoskeletal problems
* Having uncontrolled hypotension/hypertension, cardiovascular problems, metabolic and chronic diseases
* anemic individuals
* Having severe cerebrovascular and peripheral venous insufficiency
* Having had an operation in the last year

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Timed Up &Go Test | At baseline and at week 12
  This test is an assessment tool used to predict fall risk in the elderly. It is a test that measures the time between the individual getting up from the chair, walking 3 meters, and turning and sitting again. If the time taken is more than 35 seconds, it is interpreted as an increased risk of falling, while if it is less than 15 seconds, it is interpreted as a decreased risk of falling (Browne et al. 2018).
Performanz Balance System | At baseline and at week 12
  It is an electronic monitoring device designed to analyze lower extremity muscle groups that affect human balance. The basic method used is to reveal the contraction behavior of the muscles by following the balance focus. The device measured the differences between dynamic and static balance, eyes open and eyes closed balance, double leg and single leg (right/left) balance, and right/left foot balance in elderly individuals. During the test, the participant was asked to stand on the balance system and maintain his balance by following the commands given. The platform is linked to computer software that allows the balance to be evaluated objectively. Thanks to this software, measurements were monitored from the researcher's tablet or laptop (Performans Arge ve Yazılım Hizmetleri A.Ş. 2020).
Functional Reaching Test | At baseline and at week 12
  It is an easily applicable dynamic balance measurement technique that has features similar to functional movements. It is a test that can be completed in 5 minutes and evaluates how far the person can reach forward while in a fixed position and their stability during this time, accompanied by an observer. The participant is asked to stand in a stable upright position against a wall (not touching it). The arm is extended against the wall at 90 degrees and the location of the 3rd metacarpal bone is recorded. The participant is asked to lie forward as much as possible without taking a step, and the location of the 3rd metacarpal bone is recorded. The difference between the initial and final localizations of the 3rd metacarpal bone is measured. 3 trials are made and the average of the last two is taken. Distances below 15 cm have been found to be associated with an increased risk of falling (Weiner et al. 1992).
Six Minute Walking Test | At baseline and at week 12
  It is a test used to evaluate an individual's aerobic capacity. Individuals are asked to walk as much as possible for 6 minutes in a corridor that is at least 30 meters long and has a flat and hard surface. The distance traveled in 6 minutes is recorded. While the average walking distance is 570 meters for men aged 50-70 and 540 meters for women; It is stated as 530 meters for men aged 70-80 and 470 meters for women. Test results lower than these values may be associated with a decrease in aerobic capacity (American Thoracic Society 2002).
Tinetti Balance and Gait Assessment | At baseline and at week 12
  This functional test, which is used to determine the risk of falling in the elderly, contains 13 items for balance and 9 items for walking. In the balance test, each item is scored as 0, 1, 2. In the walking test, each item is scored as 0 or 1. A separate score can be calculated for balance and walking, as well as a total score. It is thought that those with scores of 26 and below have problems in terms of balance and walking functions, and it has been stated in studies that those with scores of 19 and below have a fivefold increased risk of falling compared to normal people (Tinetti 1986; Çifçili et al. 2004; Onat et al. 2014).

SECONDARY OUTCOMES:
Activity-Specific Balance and Confidence Scale | At baseline and at week 12
  It was developed by Powell and Myers to evaluate balance confidence at different levels of functions. It consists of 16 tasks related to daily living activities. A high score is associated with high confidence. Turkish validity and reliability study was conducted by Ayhan et al. (Ayhan et al. 2014).
Five Times Sit to Stand | At baseline and at week 12
  In this test, which evaluates the functional strength of the lower extremity, movement transitions, balance and risk of falling, the individual was asked to sit and stand up 5 times as fast as he could, holding his hands across his shoulders. The elapsed time was recorded with a stopwatch (Mong et al. 2010).
Montreal Cognitive Assessment Test | At baseline and at week 12
  It is an assessment scale developed to detect mild cognitive impairment. Cognitive functions evaluated in this test are attention and concentration, executive functions, memory, language, visual structuring skills, abstract thinking, calculation and orientation. It is a short and easy-to-apply scale with an application time of approximately ten minutes. The lowest score that can be obtained from the scale is 0 and the highest score is 30. A total score of 21 or above indicates that the participant is within normal limits. There are various tests used to evaluate cognitive functions in the elderly, and among these tests, the most frequently used scale is a scale that evaluates cognitive functions in different subgroups (Nasreddine et al. 2005). The Turkish validity and reliability study of the test was conducted by Ozdilek et al. (Ozdilek et al. 2014).
KATZ Activities of Daily Living Scale | At baseline and at week 12
  It is one of the most appropriate assessments to evaluate functional status as a measurement of the elderly's ability to perform daily living activities independently. Elders are scored yes/no for independence in each of six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and a score of 2 or less indicates severe functional impairment. The index, baseline measurements taken when the patient is well, is among the most effective scales used among older adults in a variety of care settings, compared to periodic or subsequent measurements (Shelkey et al. 2000). The Turkish validity and reliability study of the scale was conducted by Pehlivanoğlu et al. (Pehlivanoğlu et al. 2018).
Clinical Frailty Scale | At baseline and at week 12
  On a scale that describes the individual from 1 (Very Fit) to 9 (Terminal Illness), each category corresponds to a written description of frailty, complete with a visual chart to aid in the clinical classification of frailty. A score of ≥5 is considered mildly frail. The scale provides predictive information about length of hospital stay and mortality in older people. The validity and reliability study of the scale was conducted by Özsürekci et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Haliç University, Istanbul, Eyüpsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided